CLINICAL TRIAL: NCT04456244
Title: Comparison of Transtibial and Transfemoral Amputees' Posture Parameters
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Collaborators: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Sponsor
Other Study IDs: 19/164
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2020-06

CONDITIONS: Amputation; Traumatic, Limb; Postural; Defect
Keywords: amputation, postural adaptations, transtibial, transfemoral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:Transtibial Amputation: Photographs will be taken with posturography device during free posture and equal weighting on both extremities. Static postural adaptations will be determined by photo analysis.
  Interventions: Other: Evaluation of the static posture
- Group 2:Transfemoral Amputation: Photographs will be taken with posturography device during free posture and equal weighting on both extremities. Static postural adaptations will be determined by photo analysis.
  Interventions: Other: Evaluation of the static posture

INTERVENTIONS:
Other: Evaluation of the static posture — Photographing from the back, front and side with ADIBAS posturography in standing position

SUMMARY:
With the onset of prosthesis use following lower extremity amputations, body shows biomechanical changes according to the amputation level and consequently develops adaptation mechanisms both on the healthy and ampute side. The aim of this study is to determine the static postural adaptations that appear at different amputation levels.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having had an amputation at least 6 months ago
* Have had transfemoral amputation or transtibial amputation
* To be able to perform ambulation independently

Exclusion Criteria:

* mental inability to understand commands
* have a neurological, orthopedic and systemic problem that will negatively affect posture or gait.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — With Unilateral Transfemoral and Transtibial Amputation Patients
Study Population: With Unilateral Transfemoral and Transtibial Amputation Patients
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the static posture-1 | Changes from baseline static posture adaptations before and following Six Minutes Walking Test
  Photographing from the back, front and side with posturography (ADIBAS Posture, 1520, Kinect for XBOX ONE) in free standing position
Evaluation of the static posture-2 | Changes from baseline static posture adaptations before and following Six Minutes Walking Test
  Photographing from the back, front and side with posturography (ADIBAS Posture, 1520, Kinect for XBOX ONE) in equal weighting on platform (3D L.A.S.A.R. Posture, 743L500, Ottobock)
Evaluation of the back pain | Changes from baseline static posture adaptations before and following Six Minutes Walking Test
  Pain will be evaluated by using Visual Analog Scale ranging 0(no pain)-10(worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Kablan, PhD, Principal Investigator — Istanbul Sağlık Bilimleri Üniversitesi
Locations (1):
- Istanbul Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Silverman AK, Fey NP, Portillo A, Walden JG, Bosker G, Neptune RR. Compensatory mechanisms in below-knee amputee gait in response to increasing steady-state walking speeds. Gait Posture. 2008 Nov;28(4):602-9. doi: 10.1016/j.gaitpost.2008.04.005. Epub 2008 Jun 2. PMID 18514526
- [Result] Hendershot BD, Nussbaum MA. Persons with lower-limb amputation have impaired trunk postural control while maintaining seated balance. Gait Posture. 2013 Jul;38(3):438-42. doi: 10.1016/j.gaitpost.2013.01.008. Epub 2013 Feb 4. PMID 23391751
- [Result] Gailey R, Allen K, Castles J, Kucharik J, Roeder M. Review of secondary physical conditions associated with lower-limb amputation and long-term prosthesis use. J Rehabil Res Dev. 2008;45(1):15-29. doi: 10.1682/jrrd.2006.11.0147. PMID 18566923
- [Result] Molina-Rueda F, Alguacil-Diego IM, Cuesta-Gomez A, Iglesias-Gimenez J, Martin-Vivaldi A, Miangolarra-Page JC. Thorax, pelvis and hip pattern in the frontal plane during walking in unilateral transtibial amputees: biomechanical analysis. Braz J Phys Ther. 2014 May-Jun;18(3):252-8. doi: 10.1590/bjpt-rbf.2014.0032. PMID 25003278
- [Result] Kulkarni J, Gaine WJ, Buckley JG, Rankine JJ, Adams J. Chronic low back pain in traumatic lower limb amputees. Clin Rehabil. 2005 Jan;19(1):81-6. doi: 10.1191/0269215505cr819oa. PMID 15704512
- [Result] Soares AS, Yamaguti EY, Mochizuki L, Amadio AC, Serrao JC. Biomechanical parameters of gait among transtibial amputees: a review. Sao Paulo Med J. 2009 Sep;127(5):302-9. doi: 10.1590/s1516-31802009000500010. PMID 20169280
- [Result] Lloyd CH, Stanhope SJ, Davis IS, Royer TD. Strength asymmetry and osteoarthritis risk factors in unilateral trans-tibial, amputee gait. Gait Posture. 2010 Jul;32(3):296-300. doi: 10.1016/j.gaitpost.2010.05.003. Epub 2010 Aug 1. PMID 20678938
- [Result] Khamis S, Carmeli E. The effect of simulated leg length discrepancy on lower limb biomechanics during gait. Gait Posture. 2018 Mar;61:73-80. doi: 10.1016/j.gaitpost.2017.12.024. Epub 2017 Dec 28. PMID 29306147
- [Result] Carmona GA, Hoffmeyer P, Herrmann FR, Vaucher J, Tschopp O, Lacraz A, Vischer UM. Major lower limb amputations in the elderly observed over ten years: the role of diabetes and peripheral arterial disease. Diabetes Metab. 2005 Nov;31(5):449-54. doi: 10.1016/s1262-3636(07)70215-x. PMID 16357788
- [Result] Gaffney BM, Murray AM, Christiansen CL, Davidson BS. Identification of trunk and pelvis movement compensations in patients with transtibial amputation using angular momentum separation. Gait Posture. 2016 Mar;45:151-6. doi: 10.1016/j.gaitpost.2016.01.015. Epub 2016 Jan 25. PMID 26979898